CLINICAL TRIAL: NCT01402427
Title: Omission of Prophylactic Verapamil Use in Transradial Coronary Interventions
Brief Title: Is Verapamil In TransRadial Interventions OmittabLe?
Acronym: VITRIOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Health Center, Hungary (Other)
Responsible Party: Principal Investigator, Istvan Hizoh, MD, PhD, Senior Consultant, State Health Center, Hungary
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SHCCARD-001
Record Dates: First submitted 2011-07-21; First posted 2011-07-26 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Disease; Verapamil Toxicity
Keywords: Coronary Artery Disease; Coronary Angiography; Percutaneous Coronary Intervention; Transradial; Radial Artery Spasm; Verapamil; Adverse Effects
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Verapamil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verapamil (Active Comparator)
  Interventions: Drug: Verapamil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verapamil — Intraarterial administration of 5 mg verapamil diluted with saline to 10 mL.
  Arms: Verapamil
Drug: Placebo — Intraarterial administration of 10 mL saline.
  Arms: Placebo

SUMMARY:
Background Verapamil is traditionally applied prophylactically in transradial procedures to prevent radial artery spasm. However, verapamil may have side effects and is contraindicated in some clinical settings.

Methods: During an investigator-initiated, randomized, double-blind trial, we evaluate the need for preventive verapamil administration. After vascular access is established, patients receive either 5 mg verapamil (n=297) or placebo (n=294). We compare the rate of access site conversions as primary end point using a superiority margin of 5%. Occurrence of code breaks (composite of conversions and unplanned use of verapamil), overall verapamil use, procedural and fluoroscopic times, contrast volume, and subjective pain are investigated as secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing transradial coronary angiography and/or percutaneous coronary intervention
* successful cannulation of the radial artery

Exclusion Criteria:

* reduced left ventricular systolic function (LVEF<35%)
* significant aortic stenosis
* bradycardia (<50/min.)
* myocardial infarction complicated by cardiogenic shock and/or high grade AV block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 591 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Hizoh, MD, PhD, Principal Investigator — State Health Center, Budapest, Hungary; Robert Gabor Kiss, MD, PhD, Study Chair — State Health Center, Budapest, Hungary
Locations (1):
- State Health Center, Budapest, Hungary

REFERENCES:
- [Result] Hizoh I, Majoros Z, Major L, Gulyas Z, Szabo G, Kerecsen G, Korda A, Molnar F, Kiss RG. Need for prophylactic application of verapamil in transradial coronary procedures: a randomized trial. The VITRIOL (is Verapamil In TransRadial Interventions OmittabLe?) trial. J Am Heart Assoc. 2014 Apr 14;3(2):e000588. doi: 10.1161/JAHA.113.000588. PMID 24732918

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Verapamil | Placebo
Started | 297 | 294
Completed | 297 | 294
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Verapamil | Placebo | Total
Number analyzed (Participants) | 297 | 294 | 591
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (10.5) | 62.5 (10.8) | 62.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 104 | 215
  Male | 186 | 190 | 376
Region of Enrollment [Number; unit: participants]
  Hungary | 297 | 294 | 591

OUTCOME MEASURES:

1. Primary Outcome: Rate of Access Site Conversions
Time Frame: Occurrence of access site conversion will be assessed within 1 minute after completion of coronary angiography or intervention.
Measure: Number; unit: participants
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 297 | 294
participants | 2 | 5
Statistical Analysis 1: Comparison: Verapamil vs Placebo; Test type: Superiority or Other; p = 0.28, Fisher Exact; Risk Difference (RD) = 0.01, 95% CI 2-sided [-0.011 to 0.033]

2. Secondary Outcome: Rate of Code Breaks
Description: Code break: a composite of access site conversion and unplanned use of vasodilators.
Time Frame: Occurrence of code breaking will be assessed within 1 minute after completion of coronary angiography or intervention.
Measure: Number; unit: participants
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 297 | 294
participants | 4 | 10
Statistical Analysis 1: Comparison: Verapamil vs Placebo; Test type: Superiority or Other; p = 0.11, Fisher Exact

3. Secondary Outcome: Rate of Vasodilator Use
Time Frame: Vasodilator use will be assessed within 1 minute after completion of coronary angiography or intervention.
Measure: Number; unit: participants
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 297 | 294
participants | 297 | 6
Statistical Analysis 1: Comparison: Verapamil vs Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Procedural Time
Time Frame: Procedural time will be assessed within 1 minute after completion of coronary angiography or intervention.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 297 | 294
minutes | 17.0 [10.0 to 31.0] | 16.0 [9.0 to 30.0]
Statistical Analysis 1: Comparison: Verapamil vs Placebo; Test type: Superiority or Other; p = 0.37, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Fluoroscopic Time
Time Frame: Fluoroscopic time will be assessed within 1 minute after completion of coronary angiography or intervention.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 297 | 294
minutes | 4.8 [2.4 to 10.7] | 4.4 [2.1 to 9.6]
Statistical Analysis 1: Comparison: Verapamil vs Placebo; Test type: Superiority or Other; p = 0.28, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Contrast Volume
Time Frame: The amount of contrast medium will be assessed within 1 minute after completion of coronary angiography or intervention.
Measure: Median (Inter-Quartile Range); unit: milliliter
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 297 | 294
milliliter | 75.0 [47.0 to 156.5] | 72.5 [48.0 to 146.0]
Statistical Analysis 1: Comparison: Verapamil vs Placebo; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Subjective Pain
Description: Analysis of the rates of signiﬁcant pain deﬁned as pain score ≥4 on a semiquantitative scale ranging from 1 to 6.
Time Frame: Subjective pain will be assessed within 1 minute after completion of coronary angiography or intervention.
Measure: Number; unit: participants
Arm/Group | Verapamil | Placebo
Number analyzed (Participants) | 297 | 294
participants | 26 | 21
Statistical Analysis 1: Comparison: Verapamil vs Placebo; Test type: Superiority or Other; p = 0.45, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Verapamil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/297 | 0/294
Other Adverse Events (participants affected / at risk) | 0/297 | 0/294

LIMITATIONS AND CAVEATS:
The trial was conducted in a single, high-volume institution by experienced operators. The results may not be applicable to lower-volume centers or to operators with less experience.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes